CLINICAL TRIAL: NCT01201824
Title: Thoracoscopic Localization of Pulmonary Nodules Using Direct Intracavitary Thoracoscopic Ultrasound
Acronym: CT0007
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE 10.115
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-05

CONDITIONS: Lung Cancer
Keywords: lung cancer; intracavitary ultrasound; pulmonary nodules; VATS procedures
MeSH Terms: conditions — Lung Neoplasms; Multiple Pulmonary Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Procedure: intracavitary ultrasound

INTERVENTIONS:
Procedure: intracavitary ultrasound — intracavitary ultrasound done during surgical intervention

SUMMARY:
Pulmonary nodules are one of the most common thoracic radiographic abnormalities. They are usually found accidentally as discrete well emarginated pulmonary lesions found within the lung parenchyma during a routine chest x-ray. Pulmonary nodules are usually asymptomatic. Most solitary lung nodules are benign; however these nodules can represent early stage lung cancer. The identification of malignant pulmonary nodules is important because they represent a potential form of curable lung malignancy. Every lung nodule should therefore be investigated for the possibility of malignancy.

Ultrasound has been beneficial in almost all medical and surgical specialities. The idea of using ultrasound during VATS has emerged from its use in laparoscopic procedures. Few studies have investigated the use intracavitary ultrasound for localizing pulmonary nodules. The sensitivity of ultrasound detecting pulmonary nodules is high (92%). In some studies, ultrasound could detect all pulmonary nodules detected by high resolution CT. It has also been shown to be able to locate nodules not visualized on spiral CT.

The use of intracavitary ultrasound has been suggested by many authors as a safe and effective method for localizing hard to find nodules. It is a real time technique with no associated complications, low cost, and has the potential to save operative time. Most importantly, it may be able to prevent conversion of VATS to open operations in cases where nodules are not visualizable or locatable using VATS techniques.

The use of intracavitary US as a localization method by surgeons intra-operatively could lead to better identification of nodules. Also, this technique could avoid performing multiple procedures on patients (CT guided targeting followed by surgery) and therefore is more cost-efficient. If proven accurate, surgeon-performed intracavitary ultrasound could be used routinely during VATS procedures, increasing the chances of finding and localizing pulmonary nodules using minimally invasive techniques.

ELIGIBILITY:
Inclusion Criteria:

* All patients with CT identified pulmonary nodules not deemed to be visualizable during VATS who are candidates for VATS resection.

Exclusion Criteria:

* Inability to consent for the study.
* Patients less than 18 years old.
* Patients with pulmonary nodules easily located during VATS.
* Patients with tumours extending to visceral pleura or chest wall.
* Patients who have chest anatomy precluding VATS resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-09; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to confirm the validity of surgeon-performed intra-operative intracavitary ultrasound as a localization method for difficult to visualize pulmonary nodules during VATS procedures. | 3-6 months

SECONDARY OUTCOMES:
To assess the ability of intra-operative intracavitary ultrasound to detect new pulmonary nodules, not detected by CT. | 3-6 months
To assess the ability of VATS-US to decrease conversion rates of VATS procedures to open thoracotomy. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Monteal, Quebec, Canada

REFERENCES:
- [Derived] Khereba M, Ferraro P, Duranceau A, Martin J, Goudie E, Thiffault V, Liberman M. Thoracoscopic localization of intraparenchymal pulmonary nodules using direct intracavitary thoracoscopic ultrasonography prevents conversion of VATS procedures to thoracotomy in selected patients. J Thorac Cardiovasc Surg. 2012 Nov;144(5):1160-5. doi: 10.1016/j.jtcvs.2012.08.034. Epub 2012 Sep 12. PMID 22980667